CLINICAL TRIAL: NCT01745939
Title: The Immmediate Effects of Thrust Joint Manipulation on the Resting and Contraction Thickness of Transversus Abdominis in Subjects With Low Back Pain
Brief Title: Manipulation Effects on Abdominal Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UNLVPT-4056
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Low Back Pain
Keywords: Back pain
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar manipulation (Active Comparator): Patients will receive thrust joint manipulation to their lumbar spine in side lying
  Interventions: Other: Lumbar Manipulation
- Sham manipulation (Sham Comparator): Patients will receive oscillations into slight rotation, without cavitation, in side lying
  Interventions: Other: Sham manipulation

INTERVENTIONS:
Other: Lumbar Manipulation — Manual therapy intervention
  Arms: Lumbar manipulation
Other: Sham manipulation — Manual therapy intervention
  Arms: Sham manipulation

SUMMARY:
The purpose of this study is to understand how different physical therapy interventions affect the use of certain abdominal muscles in patients with low back pain.

DETAILED DESCRIPTION:
Patients with low back pain will undergo ultrasound imaging of the lateral abdominal wall to measure resting and contracted thickness of the transversus abdominis muscle. Following the pre-intervention measurement, patients will receive one of two physical therapy interventions (side lying thrust joint manipulation or side lying non-thrust oscillations into slight rotation) which will have been randomly assigned. Immediately after intervention, ultrasound imaging will be repeated on the resting and contracted thickness of the transversus abdominis.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving physical therapy treatment for back pain or back pain symptoms
* 18-70 years of age
* Able to perform the abdominal drawing in maneuver

Exclusion Criteria:

* Presence of a serious pathology
* Diagnosis of spinal stenosis or symptoms in both lower legs (changes in sensation, muscle weakness)
* Any history of low back surgery, rheumatoid arthritis, osteoporosis, osteopenia, or ankylosing spondylitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Transversus abdominis thickness change | Baseline to immediately after the intervention (within 5 minutes)
  Measurement of change in thickness from resting to contraction will be compared at baseline (pre-intervention) to immediately following the intervention (post-intervention). The study is looking at the immediate effects so there is no short-term or longer term follow up.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Baseline to immediately after the intervention (within 5 minutes)
  Rating of perceived pain will be compared at baseline (pre-intervention) to immediately following the intervention (post-intervention). The study is looking at the immediate effects so there is no short-term or longer term follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Durant, BSc, Study Director — University of Nevada, Las Vegas; Jade Elkind, BA, Study Director — University of Nevada, Las Vegas; Shawna Bohnet, BSc, Study Director — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas - Department of Physical Therapy, Las Vegas, Nevada, United States